CLINICAL TRIAL: NCT01977911
Title: Phase I/IIa Clinical Trial of Stem Cell Based Tissue Engineered Partial Laryngeal Implants in 10 Adult Patients With End-stage Laryngeal Stenosis With 24 Months Follow-up.
Brief Title: Clinical Trial of Stem Cell Based Tissue Engineered Laryngeal Implants
Acronym: RegenVOX
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Withdrawal of funding
Sponsor: University College, London (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL RD & ID no. 12/0331; 2013-004359-18 (EudraCT Number)
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Disorder of Upper Respiratory System; Laryngostenosis; Tracheal Stenosis
Keywords: Airway reconstruction; Regenerative medicine
MeSH Terms: conditions — Laryngostenosis; Tracheal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tissue engineered airway construct (Experimental): Stem cell based tissue engineered partial laryngeal implants:
  The final experimental product is a highly tested, recellularised, stem cells based tissue engineered product (airway construct) for operative partial laryngeal implantation into patients with severe laryngotracheal stenosis
  Interventions: Other: Stem cell based tissue engineered partial laryngeal implants

INTERVENTIONS:
Other: Stem cell based tissue engineered partial laryngeal implants — Stem cells from the patient receiving the implant are removed from the bone marrow, and are then grown on the scaffold in the laboratory. These cells will form the cartilage in the wall of the scaffold. The implant can be considered 'living' due to the cells grown on it, and this type of treatment is referred to as 'tissue engineering' or 'regenerative medicine'. Once these cells have attached and started to grow on the scaffold, it is ready to be implanted into the patient and a two separate operative stages can occur. The final stage of the operation involves removing the narrow section of voicebox or upper windpipe and implanting the scaffold to reconstruct it.
  Other Names: Tissue engineered partial laryngeal replacement graft; Tissue engineered epithelial cell layer when validated

SUMMARY:
This study aims to test a new groundbreaking treatment for narrowing of the voicebox and upper windpipe, which can be due to injury, inflammatory disease or cancer treatment. Narrowing of the voicebox or upper windpipe can leave patients dependant on a tracheostomy tube to breath through (a tube or hole in the neck), which can require a high level of care with regular hospital visits and can lead to recurrent chest infections. Regular surgical procedures may be necessary to widen the airway. Speaking may be very difficult or not even possible, breathing is usually a struggle and swallowing can also be affected. Patients feel very tired all the time.

The new treatment tested by this study is an implant that will partially replace the voicebox or upper windpipe in order to cure the narrowing. The implant is based on a human donor voicebox or windpipe that has been processed with detergents and enzymes in order to remove all the cells from the donor, leaving a 'scaffold' of connective tissue. The patient's own stem cells are removed from the bone marrow, then are grown on the scaffold in the laboratory. These cells will form the cartilage in the wall of the scaffold. A split skin graft from the patient may be needed to line the inside of the implant. The implant can be considered 'living' due to the cells grown on it, and this type of treatment is referred to as 'tissue engineering' or 'regenerative medicine'.

Once these cells have attached and started to grow on the scaffold, it is ready to be implanted into the patient, and an operation is performed which occurs in two separate stages. The final stage of the operation involves removing the narrow section of voicebox or upper windpipe and implanting the scaffold to reconstruct it. Patients will be followed up for two years after this operation, with investigations such as CT scans, examination of the voicebox and windpipe with a flexible camera (bronchoscopy) and blood tests performed at specific times.

It is intended that this treatment will significantly improve patients' symptoms resulting in better breathing, swallowing and voice function, reducing the need for repeated hospital visits and procedures and enhancing patients' quality of life.

DETAILED DESCRIPTION:
The RegenVOX trial is a phase I/IIa safety and potential efficacy clinical trial of tissue-engineered laryngotracheal replacement using autologous-derived cells and decellularised human donor scaffolds in 10 patients with severe acquired laryngotracheal stenosis.

Current solutions for the treatment of advanced structural disorders of the larynx such as trauma, inflammatory disorders or following cancer treatment are suboptimal and patients with such problems require frequent hospitalisation. A regenerative solution that restores the anatomy of the larynx would provide a definitive treatment for these patients, improve the outcome of resection for malignant disease, avoid some laryngectomies and would reduce the threshold for performing surgery over administering chemotherapy thereby reducing morbidity. Giving patients a once-only therapy of a life-time functional living replacement would allow patients to lead tracheostomy-free lives with improved breathing, swallowing and speech and a lower requirement for hospital follow-up.

This project is a clinical trial of tissue engineered partial laryngeal replacements in 10 patients with end-stage laryngeal stenosis. The intervention is based on a human donor graft scaffold which is decellularised and then seeded with autologous mesenchymal stem cell-derived chondrocytes externally. Following expansion of these cells ex-vivo, the graft is implanted. This is the first clinical trial to our knowledge of a stem-call based organ replacement.

Inclusion criteria are:

Patients aged >=18 years with sufficient numbers of Mesenchymal Stromal Cells (MSCs) in their human Bone Marrow (hBM) aspirate.

Patients with Myer-Cotton Grade 3 or 4 laryngotracheal stenosis or malacia due to traumatic, inflammatory, iatrogenic, or idiopathic causes who have exhausted conventional therapies.

Exclusion criteria are:

Pregnancy. Patients positive for HIV 1, HIV 2, Hepatitis C (HCV), Hepatitis B (HBV), syphilis or Human T-cell Lymphotropic Virus (HTLV).

Those unable to provide informed consent. Co-morbid severe chronic obstructive pulmonary disease (according to NICE criteria) Patients with active / uncontrolled chronic inflammatory conditions such as granulomatosis with polyangitis (formerly Wegener's granulomatosis) and sarcoidosis.

Any current or previous cancer within 5 years (except non-melanoma skin cancer, adequately treated carcinoma in situ of the uterine cervix, laryngeal malignancy treated locally with no local recurrence and no metastases, or low grade airway malignancy such as chondrosarcoma which may be causing airway obstruction).

Life expectancy less than 5 years unless this limitation is principally due to the airway obstruction to be treated.

Concurrent enrollment in any other Clinical Trial of Investigational Medicinal Product (CTIMP).

The primary outcome measure is safety as determined by morbidity and mortality as measured by occurrence of adverse events. Secondary outcome is efficacy as determined by

1. Absence of tracheostomy.
2. Absence of non-absorbable stent.
3. Improvement in mean airway diameter.
4. Improvement in Forced Expiratory Volume in 1 second (FEV1).
5. Improvement in global quality of life (EQ-5D).
6. Improvement in maximum phonation time (MPT) as measured by Voice Analysis Operavox (VAO).
7. Improvement in self assessment of voice handicap (VHI-10).
8. Improvement in swallowing function (EAT-10).
9. Improvement in airway, dyspnoea, voice, swallowing index (ADVS index).
10. Improvement in the penetration-aspiration scale (PAS) as per Video Fluoroscopic Swallow (VFS) or Functional Endoscopic Evaluation of Swallowing (FEES).

Health economics. Patients will be followed up for 2 years within this study. Key milestones will be assessed at 6 and 12 months. The follow-up regimen includes bronchoscopy and airway brushings taken at 1 week post implantation and full physical assessment including CT imaging, pulmonary function tests, blood tests and bronchoscopy at 1, 6, 12, 18 and 24 months. Telephone follow-up will take place in between these assessments.

This trial will provide a level of insight into the real clinical potential for stem cell/tissue engineering combined technologies. The results will have wide implications for the development of hollow organ- replacements such as those for oesophagus, bowel and vascular disorders. We will also develop new pathways for maximising discovery science and health economic benefit from complex regenerative medicine therapies (a reverse translational route map), with important generic benefits for scientists and clinicians.

ELIGIBILITY:
Inclusion Criteria:

Patients aged >=18 years with sufficient numbers of Mesenchymal Stromal Cells (MSCs) in their 8-10ml human Bone Marrow (hBM) aspirate.

Patients with Myer-Cotton Grade 3 or 4* laryngotracheal stenosis or equivalent due to traumatic, inflammatory, iatrogenic, or idiopathic causes who have exhausted conventional therapies.

*The Myer-Cotton grading system for mature, firm, circumferential stenosis, confined to the subglottis describes the stenosis based on the per cent relative reduction in cross-sectional area of the subglottis. Four grades of stenosis:

* grade 1 lesions have less than 50% obstruction
* grade 2 lesions have 51% to 70% obstruction
* grade 3 lesions have 71% to 99% obstruction
* grade 4 lesions have no detectable lumen or complete stenosis

Exclusion Criteria:

* Pregnancy
* Patients positive for HIV 1, HIV 2, HCV, HBV, syphilis or HTLV
* Those unable to provide informed consent
* Co-morbid severe chronic obstructive pulmonary disease (according to NICE criteria)
* Patients with active / uncontrolled chronic inflammatory conditions such as granulomatosis with polyangitis (formerly Wegener's granulomatosis) and sarcoidosis
* Any current or previous cancer within 5 years (except non-melanoma skin cancer, adequately treated carcinoma in situ of the uterine cervix, laryngeal malignancy treated locally with no local recurrence and no metastases, or low grade airway malignancy such as chondrosarcoma which may be causing airway obstruction)
* Life expectancy less than 5 years unless this limitation is principally due to the airway obstruction to be treated
* Concurrent enrollment in any other Clinical Trial of Investigational Medicinal Product (CTIMP).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04 (Estimated); Primary Completion 2018-05-25 (Actual); Study Completion 2018-05-25 (Actual)

PRIMARY OUTCOMES:
Safety of tissue engineered laryngotracheal replacement | 24 months post operative follow up
  The primary outcome measure is safety of the tissue engineered implant as defined by morbidity and mortality and measured by occurrence of adverse events throughout 24 months post operative follow up

SECONDARY OUTCOMES:
Efficacy of tissue engineered laryngotracheal replacement | 24 months post operative follow up
  Secondary outcome is efficacy as determined
  1. Absence of tracheostomy.
  2. Absence of non-absorbable stent.
  3. Improvement in mean airway diameter.
  4. Improvement in Forced Expiratory Volume in 1 second (FEV1).
  5. Improvement in global quality of life (EQ-5D).
  6. Improvement in maximum phonation time (MPT) as measured by Voice Analysis Operavox (VAO).
  7. Improvement in self assessment of voice handicap (VHI-10).
  8. Improvement in swallowing function (EAT-10).
  9. Improvement in airway, dyspnoea, voice, swallowing index (ADVS index).
  10. Improvement in the penetration-aspiration scale (PAS) as per Video Fluoroscopic Swallow (VFS) or Functional Endoscopic Evaluation of Swallowing (FEES).
  Health Economics

OTHER OUTCOMES:
Cost effectiveness of tissue engineered laryngotracheal replacement | 24 months post operative follow up
  We will also develop new pathways for maximising discovery science and health economic benefit from complex regenerative medicine therapies (a reverse translational route map), with important generic benefits for scientists and clinicians.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Birchall, Prof, Principal Investigator — University College London (UCL) Ear Institute; Royal National Throat, Nose and Ear Hospital
Locations (1):
- University College London NHS Foundation Trust (UCLH), London, United Kingdom

REFERENCES:
- [Background] Hamilton N, Bullock AJ, Macneil S, Janes SM, Birchall M. Tissue engineering airway mucosa: a systematic review. Laryngoscope. 2014 Apr;124(4):961-8. doi: 10.1002/lary.24469. Epub 2013 Nov 19. PMID 24129819
- [Derived] Culme-Seymour EJ, Mason K, Vallejo-Torres L, Carvalho C, Partington L, Crowley C, Hamilton NJ, Toll EC, Butler CR, Elliott MJ, Birchall MA, Lowdell MW, Mason C. Cost of Stem Cell-Based Tissue-Engineered Airway Transplants in the United Kingdom: Case Series. Tissue Eng Part A. 2016 Feb;22(3-4):208-13. doi: 10.1089/ten.TEA.2015.0283. Epub 2015 Dec 24. PMID 26559535
- See also: Related systematic review; PMID 24129819 [doi] full text — http://onlinelibrary.wiley.com/doi/10.1002/lary.24469/abstract;jsessionid=1C529728C706053B92F089E7EB999046.f02t01